CLINICAL TRIAL: NCT03852537
Title: SMART Trial: Steroid Dosing by bioMARker Guided Titration in Critically Ill Patients With Pneumonia
Brief Title: Steroid Dosing by bioMARker Guided Titration in Critically Ill Patients With Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hemang Yadav, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-010925
Record Dates: First submitted 2019-02-15; First posted 2019-02-25 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pneumonia
Keywords: Pneumonia, steroid, COVID-19, SARS CoV-2
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Usual care as determined by the patient's primary team.
  Interventions: Other: Usual Care
- Biomarker-adjusted Steroid Dosing (Experimental): Individualized, biomarker concordant steroid use: dosing, titration and duration according to CRP level. This is a predetermined dosing table that adjusts dose of steroid by CRP level. Specifically: if CRP < 50 mmol/L: discontinue steroid; if CRP is between 51-100 mmol/L: 0.5 mg methylprednisolone (or dose equivalent of oral prednisone); if CRP is between 101-150 mmol/L: 0.75 mg/kg methylprednisolone (or dose equivalent of oral prednisone); if CRP level is between 151-200 mmol/L: 1 mg/kg methylprednisolone (or dose equivalent of oral prednisone); if CRP level > 200 mmol/L: 1.5 mg/kg methylprednisolone (or dose equivalent of oral prednisone).
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone will be administered based on CRP-guided protocol outlined under 'Biomarker-adjusted steroid dosing'.
  Other Names: Biomarker guided steroid dosing
  Arms: Biomarker-adjusted Steroid Dosing
Other: Usual Care — Usual care as determined by the patients treatment team.
  Arms: Usual Care

SUMMARY:
This research study is being done to determine the appropriate dose of steroids and the appropriate duration for steroid use to reduce inflammation in severe pneumonia needing a form of breathing support. This study seeks to compare usual care to a unique (individualized) dosing strategy. A marker of inflammation in the body will be measured in blood samples. This marker of inflammation is called C- reactive protein. The overall goal is to identify patients that will benefit most from steroid use and decrease use of steroids. The information collected from this study may provide information that may improve management of patients with severe pneumonia requiring a form of breathing support.

DETAILED DESCRIPTION:
This is a two-arm single-center pilot phase II clinical trial. Patients will be screened at the time of hospital admission and will be required to be enrolled within the clinical trial within 48 hours of hospital admission.

In the individualized, biomarker-concordant arm, all patients will receive steroids once at the time of admission, then a daily morning dose. In order to account for varying turnaround time at different laboratories, C-Reactive Protein (CRP) levels will be drawn with early morning labs, and used to determine the steroid dosing for the day. Patients will receive daily CRP measurements for the first 5 days of the hospitalization, or until hospital discharge. CRP measurements will be discontinued once the CRP is less than 50mmol/L.

Steroid administration will be facilitated using standardized computerized physician order entry. The patients, treating physicians and outcome assessors will be blinded to the group assignment. Steroid order sets will include 6 hourly point of care glucose monitoring, and an insulin sliding scale for glucose levels to facilitate glucose management. The need for insulin drip will be determined by the treating physician. Additional testing including serum and urine ketones will be informed by the glucose level, serum anion gap and bicarbonate levels in routine basic metabolic panels and determined by the treating physician.

In the usual care arm, patients will receive daily CRP measurements for the first 5 days of the hospitalization, or until hospital discharge.

ELIGIBILITY:
For the Pneumonia arm of the study:

Inclusion Criteria:

* Patients admitted to hospital with community acquired pneumonia.
* Acute respiratory failure SpO2/FiO2 < 315 (SpO2<90% on room air or <97% on 2L NC).

Exclusion Criteria:

* Contraindications or unwilling to use steroids by patient or provider
* Refractory septic shock defined as a requirement of norepinephrine dose or equivalent above >0.1 microgram/kilogram/minute or 2 or more vasopressors
* Pre-admission chronic use of steroids or other immunosuppressive medications
* Adrenal insufficiency
* Comfort care
* Leukopenia <1000/mm or neutropenia <500/mm (except if attributable to pneumonia) and HIV positive with a CD4 count <100
* Recent or past history of bone marrow or solid organ transplantation
* Hospital admission in the previous 30 days
* Suspected flare of Interstitial lung disease (infectious and non-infectious)
* Positive influenza testing or high suspicion for influenza

For the COVID-19 arm of the study:

Inclusion Criteria:

* Patients admitted to hospital with COVID-19 pneumonia (high suspicion or confirmed by positive SARS CoV-2 testing).
* Acute respiratory failure SpO2/FiO2 < 315 (SpO2<90% on room air or <97% on 2L NC).

Exclusion Criteria:

* Contraindications or unwilling to use steroids by patient or provider
* Refractory septic shock defined as a requirement of norepinephrine dose or equivalent above >0.1 microgram/kilogram/minute or 2 or more vasopressors
* Pre-admission chronic use of steroids or other immunosuppressive medications
* Adrenal insufficiency
* Comfort care
* Leukopenia <1000/mm or neutropenia <500/mm (except if attributable to pneumonia) and HIV positive with a CD4 count <100
* Recent or past history of bone marrow or solid organ transplantation
* Suspected flare of Interstitial lung disease (infectious and non-infectious)
* Positive influenza testing or high suspicion for influenza

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hemang Yadav, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any manuscript resulting from this research, after deidentification (text, tables, figures, and appendices) and the study protocol will be shared beginning 9 months and ending 36 months following article publication, to anyone who wishes to access the data. Proposals should be directed to yadav.hemang@mayo.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 9 months to 36 months after article publication.

REFERENCES:
- [Derived] Odeyemi YE, Chalmers SJ, Barreto EF, Jentzer JC, Gajic O, Yadav H. Early, biomarker-guided steroid dosing in COVID-19 Pneumonia: a pilot randomized controlled trial. Crit Care. 2022 Jan 4;26(1):9. doi: 10.1186/s13054-021-03873-2. PMID 34983600
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Corticosteroid use and dosing determined by the patient's primary team for standard of care.
  Usual Care: Corticosteroid use and dosing determined by the patients treatment team for standard of care.
Period: Overall Study
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [50.0 to 67.0] | 59.0 [52.0 to 79.0] | 60.0 [51.5 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Timely Initiation of Corticosteroids and Implementation of Biomarker-titrated Corticosteroid Dosing
Description: Number of eligible subjects to adhered to the timely initiation and daily corticosteroid treatment according to ESICM/Society of Critical Care Medicine SCCM clinical practice guideline (control group) or biomarker concordance (intervention group)
Time Frame: Within 30 days of enrollment in study.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 20 | 19

2. Secondary Outcome: Mortality
Description: Number of subject deaths
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 1 | 1

3. Secondary Outcome: Need for High Flow Nasal Cannula Oxygen
Description: Number of subjects to need high flow nasal cannula oxygen
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 7 | 4
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 0.494, Fisher Exact

4. Secondary Outcome: Need for Noninvasive Mechanical Ventilation
Description: Assessed by the number of participants that required noninvasive mechanical ventilation.
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 4 | 2
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 0.666, Fisher Exact

5. Secondary Outcome: Need for Invasive Mechanical Ventilation
Description: Assessed by the number of participants that required invasive mechanical ventilation.
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 3 | 2
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 1.000, Fisher Exact

6. Secondary Outcome: Organ Failure
Description: Organ failures measured by Sequential Organ Failure Assessment (SOFA). The overall score is based on 6 sub-scores respiratory system, neurologic system, cardiovascular system, hepatic system, coagulation, and renal system using an overall scale of 0-24, which 0=no organ failure, 24=complete organ failure.
Time Frame: Measured daily for approximately 5 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
score on a scale
  Day 1 | 3.0 [3.0 to 6.0] | 7.0 [4.0 to 9.0]
  Day 2 | 3.0 [3.0 to 3.0] | 3.0 [2.0 to 6.0]
  Day 3 | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 5.5]
  Day 4 | 3.0 [3.0 to 5.0] | 3.0 [2.0 to 8.0]
  Day 5 | 3.0 [2.0 to 5.0] | 5.5 [3.0 to 8.0]

7. Secondary Outcome: New Onset Cardiac Arrhythmias
Description: Number of participants who develop arrhythmias identified by electrocardiogram or echocardiogram.
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 0 | 1
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 0.477, Fisher Exact

8. Secondary Outcome: Myocardial Injury
Description: Number of participants with evidence of myocardial injury determined by daily troponin peak and /or new diagnosis of Left Ventricular (LV) dysfunction (LVEF <40%) or new diagnosis of cor pulmonale
Time Frame: Up to day +14 following study enrollment.
Population: Data were missing for 8 subjects in the usual care arm and 4 subjects in the biomarker-adjusted steroid dosing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 15 | 17
Participants | 8 | 10
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 1.000, Chi-squared

9. Secondary Outcome: Cardiovascular Dysfunction
Description: Number of subjects with new and/or worsening right ventricle (RV)/left ventricle (LV) dysfunction
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 1 | 1
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 1.000, Fisher Exact

10. Secondary Outcome: Occurrence of Hyperglycemia
Description: Number of participants who have hyperglycemia while receiving corticosteroids. Hyperglycemia is defined as a consistently elevated blood sugar level requiring insulin administration.
Time Frame: Up to day +5 following study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 11 | 18
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 0.011, Fisher Exact

11. Secondary Outcome: Occurrence of Delirium
Description: Number of participants who develop delirium while receiving corticosteroids. Delirium will be assessed by Confusion Assessment Method for the ICU (CAM-ICU) measurement tool. The CAM-ICU is a binary (yes/no) scale for assessing the presence of delirium.
Time Frame: Up to day +5 following study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 5 | 5
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 1.000, Fisher Exact

12. Secondary Outcome: Occurrence of Secondary Infection
Description: Number of participants who develop secondary infections during and after steroid therapy. A secondary infection is defined as a new infection that develops after initiation of corticosteroid therapy, until 5 days after steroids are discontinued.
Time Frame: Up to day +14 following study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 0 | 0

13. Secondary Outcome: ICU Admission
Description: Number of subjects admitted to the ICU
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
Participants | 10 | 5
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-adjusted Steroid Dosing; Test type: Superiority; p = 0.213, Chi-squared

14. Secondary Outcome: Oxygen-free Days
Description: Number of days subjects did not require oxygen assistance.
Time Frame: Within hospitalization or 30 days of study enrollment (whichever is sooner)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
Number analyzed (Participants) | 23 | 21
days | 21.0 [17.0 to 25.0] | 24.0 [22.0 to 25.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 90 days on all participants.
Arm/Group | Usual Care | Biomarker-adjusted Steroid Dosing
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03852537/Prot_SAP_000.pdf